CLINICAL TRIAL: NCT05574478
Title: Evaluation of the Acceptability, Appropriateness, Feasibility and Utility of a Metastatic Breast Cancer-Specific Prognostic Tool Among Patients With Metastatic Breast Cancer and Their Caregivers
Brief Title: Metastatic Breast Cancer-Specific Prognostic Tool
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Conquer Cancer Foundation (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2213
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Patients; End of life; Caregivers
MeSH Terms: conditions — Breast Neoplasms; Death

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients and Caregivers: Participants will include patients diagnosed with metastatic breast cancer and caregivers for patients diagnosed with metastatic breast cancer. Participants will be recruited from the UNC Medical Center breast oncology group as well as other practices identified by the Principal Investigator based on existing professional networks (referring physicians, other UNC oncology entities, collaborative groups).
  Interventions: Behavioral: Patients and Caregivers Qualitative Interview

INTERVENTIONS:
Behavioral: Patients and Caregivers Qualitative Interview — Interviews will be conducted by experienced qualitative researchers from the UNC Connected Health for Applications & Interventions (CHAI) Core. The interview will be conducted over the phone or secure videoconferencing. The interview will be conducted in a semi-structured fashion using an interview guide. However, because the purpose of this semi-structured qualitative interview study is to determine which themes participants identify as important, the exact content of each interview will differ, and the interview guide will be modified as additional interviews are conducted. Interviews will be audio recorded with concurrent notetaking by the interviewer.

SUMMARY:
In this qualitative study, Investigators will conduct semi-structured interviews with clinicians that are involved in the care of patients with breast cancer to evaluate the acceptability, appropriateness, and feasibility/usability of a metastatic breast cancer-specific prognostic tool. These interviews will be conducted by the UNC CHAI Core and will continue until thematic saturation (estimated 20-30 participants). The investigators will code the qualitative data using emerging themes, guided by a well-established implementation science theory, the Consolidated Framework for Implementation Research (CFIR). The information gained from these studies will inform an implementation approach to increase the usability and acceptability of a novel prognostic tool to assist oncologists in the prognosis of patients with metastatic breast cancer.

DETAILED DESCRIPTION:
If this study is successful, Investigators will implement an MBC-specific prognostic tool to help clinicians identify patients who are at high risk of death in the next 30 days. Based on the input from clinicians in this proposal, as well as additional qualitative studies with patients and families, Investigators will design an implementation protocol to inform how to use this tool in clinical practice. Rather than simply publishing a prognostic tool that may not be adopted into practice, this project aims to ensure successful implementation of an evidence-based tool into the routine care of patients with MBC. Doing so will serve as an important step towards identifying high-risk patients and connecting ort to ensure high-quality, patient-centered end-of-life care.

ELIGIBILITY:
Inclusion Criteria:

1. In order to participate in this study a subject must meet ALL of the eligibility criteria outlined below.
2. Subjects is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
3. Diagnosis of metastatic breast cancer or primary caregiver for someone with a diagnosis of metastatic breast cancer
4. Age > 18 years
5. Verbal informed consent obtained to participate in the study.
6. Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

Exclusion Criteria:

1. Non-English speaking

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients diagnosed with metastatic breast cancer and/or caregivers of patients diagnosed with metastatic breast cancer. Participants will be recruited from the UNC Medical Center breast oncology group as well as other practices identified by the Principal Investigator based on existing professional networks (referring physicians, other UNC oncology entities, collaborative groups).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Determining the key patient and caregiver factors impacting implementation of a metastatic breast cancer prognostic tool through semi-structured qualitative interviews. | 12 months
  Study Investigators have developed a metastatic breast cancer (MBC)-specific prognostic calculator using the ASCO CancerLinQ Discovery database to help oncologists better estimate prognosis in MBC patients. Key factors impacting implementation of a MBC prognostic tool will be evaluated through semi-structured qualitative interviews with patients and caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Ray, MD, Principal Investigator — University of North Carolina
Locations (1):
- Terri Eubanks, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials